CLINICAL TRIAL: NCT00515151
Title: Skin Disinfection With Octenidine Dihydrochloride for the Prevention of Catheter-Associated Infections - A Double-Blind, Randomized, Controlled Trial
Brief Title: Prevention of Catheter-Associated Infection With the Skin Disinfectant Octenidine Dihydrochloride
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Collaborators: University Hospital, Basel, Switzerland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NEO-0102
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Last update posted 2007-08-13 (Estimated); Status verified 2007-08

CONDITIONS: Catheterization, Central Venous; Catheter-Associated Infections; Bacterial Infections; Bacteremia
Keywords: Bloodstream Infection; Bacteremia; Central Venous Catheter; Alcohol; Disinfection; Octenidine Dihydrochloride
MeSH Terms: conditions — Catheter-Related Infections; Bacterial Infections; Bacteremia; Sepsis | interventions — octenidine; 1-Propanol; 2-Propanol; Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oct/Alc (Active Comparator)
  Interventions: Drug: 0.1% Octenidine with 30% 1-propanol and 45% 2-propanol
- Alc (Active Comparator)
  Interventions: Drug: 74% Ethanol with 10% 2-propanol

INTERVENTIONS:
Drug: 0.1% Octenidine with 30% 1-propanol and 45% 2-propanol — Before insertion of the catheter, the entry site was disinfected with the assigned solution over an area of >200 cm² for at least one minute. The assigned solution was then applied for care of the entry site during the change of dressings, usually every 2 to 3 days.
  Other Names: Octeniderm; Neo-Kodan
  Arms: Oct/Alc
Drug: 74% Ethanol with 10% 2-propanol — Before insertion of the catheter, the entry site was disinfected with the assigned solution over an area of >200 cm² for at least one minute. The assigned solution was then applied for care of the entry site during the change of dressings, usually every 2 to 3 days.
  Other Names: Softasept
  Arms: Alc

SUMMARY:
Health-care-acquired infections are of tremendous importance for patients, especially catheter-associated infections. More than 40% of all bloodstream infections are associated with central venous catheters (CVC; catheters which are inserted into a large vein near the heart). Of all patients that acquire such an infection 1% to 5% die as a result from it. The insertion site is the main source of contamination and infection. In general, bacteria of the skin are the cause of infection, especially in short-term CVCs (10-14 days). Therefore it is necessary to efficiently disinfect the skin for the preparation and care of CVC insertion sites. Several substances are used for disinfection. Alcohol-based disinfectants are mainly used in Central Europe, other preparations contain povidine-iodine or chlorhexidine. Alcoholic disinfectants have a rapid initial effect, chlorhexidine shows an additional remanent (longer lasting) effect. A further substance, octenidine dihydrochloride, also demonstrated a remanent effect in a pilot study with neurosurgical patients. The purpose of our study is to compare an alcohol-based disinfectant containing octenidine dihydrochloride with a pure alcoholic disinfectant regarding efficacy and tolerability in patients receiving a CVC for a minimum of 5 days.

DETAILED DESCRIPTION:
Catheter-associated infections are one of the most eminent healthcare acquired infections. More than 40% of all bloodstream infections are associated with a central venous catheter (CVC)and between 1% and 5% of the affected patients die as a direct consequence of this infection. The most important microorganisms are gram-positive cocci (S. aureus, S. epidermidis). In intensive care units gram-negative microorganisms such as pseudomonas, acinetobacter and candida spp. are more frequent. The insertion site is the main source of contamination and infection in short-term CVCs (10-14 days. In this case the infection is caused by migration of microorganisms along the outside of the catheter. Contamination of the hub due to frequent manipulation is usually the source of infection in long-term CVCs. In this case the infection occurs intraluminally. An effective skin disinfection is the main measure of prevention before insertion of a CVC. The aim of this measure is the elimination of transient and the reduction of resident microorganisms around the insertion site. To achieve this, disinfectants on the basis of alcohol, povidone-iodine or chlorhexidine are applied. Alcohol-based disinfectants are preferred in Central Europe because of their rapid initial effect and broad microbiological spectrum. Chlorhexidine and povidone-Iodine in contrast to alcoholic disinfectants have a remanent effect which reduces regrowth of microorganisms beyond the immediate initial effect. To which extent remanent substances reduce colonization of the CVC extraluminally or the CVC-tip is still being disputed. In an earlier clinical trial a residual or remanent effect of 0.1% octenidine combined with propanol in microbial skin decontamination over a 24h period was shown in neurosurgical patients receiving a central line (CVC or peripherally inserted central catheter). The objective of this study is therefore to evaluate further the preventive impact and tolerability of a commercially available, alcohol-based antiseptic solution containing octenidine for the preparation and care of CVC insertion sites in a clinical setting in comparison with the results given by an alcoholic solution alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years
* Medical indication for CVC with a planned duration of minimum 5 days
* Patient´s (or relative´s if applicable) written informed consent

Exclusion Criteria:

* Known sensitisation against the proposed antiseptics
* Tunneled or implanted CVCs (e.g. Hickman Catheter)
* Administration of antimicrobial drugs for therapy (not prophylaxis) less than one week prior to catheterization
* Pre-existing bloodstream infection (i.e., fever and/or other signs of infection)
* Positive blood culture
* Terminal patients with limited therapy options
* Patients with burns
* Patients participating in a clinical trial on other antiseptics within a period of four weeks prior to inclusion date
* Patients with missing written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2002-05; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Skin colonisation in cfu/cm2 at the insertion site; Colonisation of the CVC-tip, positivity by definition of number cfu/5cm > 15 (Maki-method); Incidence of catheter-associated bloodstream infection | For the duration of catheter placement plus 2 days

SECONDARY OUTCOMES:
Comparison of therapy regimens regarding side effects and complications | For the duration of catheter placement plus 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Markus Dettenkofer, Prof. MD, Principal Investigator — Institute of Environmental Medicine and Hospital Epidemiology University Medical Center Freiburg, Germany
Locations (2):
- Institute of Environmental Medicine and Hospital Epidemiology University Medical Center Freiburg, Freiburg im Breisgau, Germany
- Division of Infectious Diseases and Hospital Epidemiology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Background] Mermel LA. Prevention of intravascular catheter-related infections. Ann Intern Med. 2000 Mar 7;132(5):391-402. doi: 10.7326/0003-4819-132-5-200003070-00009. PMID 10691590
- [Background] Dettenkofer M, Wenzler-Rottele S, Babikir R, Bertz H, Ebner W, Meyer E, Ruden H, Gastmeier P, Daschner FD; Hospital Infection Surveillance System for Patients with Hematologic/Oncologic Malignancies Study Group. Surveillance of nosocomial sepsis and pneumonia in patients with a bone marrow or peripheral blood stem cell transplant: a multicenter project. Clin Infect Dis. 2005 Apr 1;40(7):926-31. doi: 10.1086/428046. Epub 2005 Mar 4. PMID 15824981
- [Background] Raad I. Intravascular-catheter-related infections. Lancet. 1998 Mar 21;351(9106):893-8. doi: 10.1016/S0140-6736(97)10006-X. No abstract available. PMID 9525387
- [Background] Safdar N, Maki DG. The pathogenesis of catheter-related bloodstream infection with noncuffed short-term central venous catheters. Intensive Care Med. 2004 Jan;30(1):62-7. doi: 10.1007/s00134-003-2045-z. Epub 2003 Nov 26. PMID 14647886
- [Background] O'Grady NP, Alexander M, Dellinger EP, Gerberding JL, Heard SO, Maki DG, Masur H, McCormick RD, Mermel LA, Pearson ML, Raad II, Randolph A, Weinstein RA; Healthcare Infection Control Practices Advisory Committee. Guidelines for the prevention of intravascular catheter-related infections. Infect Control Hosp Epidemiol. 2002 Dec;23(12):759-69. doi: 10.1086/502007. PMID 12517020
- [Background] Chaiyakunapruk N, Veenstra DL, Lipsky BA, Saint S. Chlorhexidine compared with povidone-iodine solution for vascular catheter-site care: a meta-analysis. Ann Intern Med. 2002 Jun 4;136(11):792-801. doi: 10.7326/0003-4819-136-11-200206040-00007. PMID 12044127
- [Background] Sedlock DM, Bailey DM. Microbicidal activity of octenidine hydrochloride, a new alkanediylbis[pyridine] germicidal agent. Antimicrob Agents Chemother. 1985 Dec;28(6):786-90. doi: 10.1128/AAC.28.6.786. PMID 3909955
- [Background] Buhrer C, Bahr S, Siebert J, Wettstein R, Geffers C, Obladen M. Use of 2% 2-phenoxyethanol and 0.1% octenidine as antiseptic in premature newborn infants of 23-26 weeks gestation. J Hosp Infect. 2002 Aug;51(4):305-7. doi: 10.1053/jhin.2002.1249. PMID 12183146
- [Background] Tietz A, Frei R, Dangel M, Bolliger D, Passweg JR, Gratwohl A, Widmer AE. Octenidine hydrochloride for the care of central venous catheter insertion sites in severely immunocompromised patients. Infect Control Hosp Epidemiol. 2005 Aug;26(8):703-7. doi: 10.1086/502606. PMID 16156327
- [Background] Dettenkofer M, Jonas D, Wiechmann C, Rossner R, Frank U, Zentner J, Daschner FD. Effect of skin disinfection with octenidine dihydrochloride on insertion site colonization of intravascular catheters. Infection. 2002 Oct;30(5):282-5. doi: 10.1007/s15010-002-2182-2. PMID 12382087
- [Background] Bouza E, Alvarado N, Alcala L, Sanchez-Conde M, Perez MJ, Munoz P, Martin-Rabadan P, Rodriguez-Creixems M. A prospective, randomized, and comparative study of 3 different methods for the diagnosis of intravascular catheter colonization. Clin Infect Dis. 2005 Apr 15;40(8):1096-100. doi: 10.1086/428576. Epub 2005 Mar 17. PMID 15791507
- [Background] Eggimann P, Harbarth S, Constantin MN, Touveneau S, Chevrolet JC, Pittet D. Impact of a prevention strategy targeted at vascular-access care on incidence of infections acquired in intensive care. Lancet. 2000 May 27;355(9218):1864-8. doi: 10.1016/S0140-6736(00)02291-1. PMID 10866442
- [Background] Maki DG, Ringer M, Alvarado CJ. Prospective randomised trial of povidone-iodine, alcohol, and chlorhexidine for prevention of infection associated with central venous and arterial catheters. Lancet. 1991 Aug 10;338(8763):339-43. doi: 10.1016/0140-6736(91)90479-9. PMID 1677698
- [Derived] Dettenkofer M, Wilson C, Gratwohl A, Schmoor C, Bertz H, Frei R, Heim D, Luft D, Schulz S, Widmer AF. Skin disinfection with octenidine dihydrochloride for central venous catheter site care: a double-blind, randomized, controlled trial. Clin Microbiol Infect. 2010 Jun;16(6):600-6. doi: 10.1111/j.1469-0691.2009.02917.x. Epub 2009 Aug 17. PMID 19686276